CLINICAL TRIAL: NCT01055392
Title: Disease-modifying Properties of Lithium in the Neurobiology of Alzheimer's Disease: a Double-blind, Placebo-controlled Prevention Study in Elderly Patients With Mild Cognitive Impairment
Brief Title: Disease-modifying Properties of Lithium in the Neurobiology of Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Orestes Vicente Forlenza, Department and Institute of psychiatry, Faculty of Medicine - University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OVForlenza-Lithium; 554535/2005-0 (Other Grant/Funding Number: Conselho Nacional de Pesquisa Científica)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2009-12

CONDITIONS: Cognitive Impairment; Alzheimer Disease
Keywords: mild cognitive impairment; Alzheimer's disease; Lithium; disease-modification; cognition; early Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lithium (Experimental): Patients received low doses of lithium salts (from 150 mg to 450 mg of lithium salts daily) to achieve sub-therapeutic lithium levels (target serum lithium level of 0,25 - 0,5 mEq/L). Lithium doses were administered twice a day. Lithium doses were titrated to achieve the target serum lithium levels within the first two weeks after study recruitment. After achieving the target serum lithium level, lithium salts doses remained stable until the end of the study.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Identical placebo tablets were administered twice-a-day for two years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — lithium carbonate tablets, 150 mg to 450 mg (target serum lithium level 0.25 mEq/L - 0.5 mEq/L), divided in two doses, two years.
  Arms: Lithium
Drug: Placebo — Identical placebo tablets were administered twice-a-day for two years.
  Arms: Placebo

SUMMARY:
Lithium salts have been used for the treatment of psychiatric disorders for over five decades, mostly as a mood-stabilizing drug. Recent evidence points to the inhibition of the enzyme glycogen synthase kinase-3beta (GSK3) as one of its mechanisms of action. The overactivity of this enzyme has been implicated in the pathogenesis of Alzheimer's disease (AD), given its involvement in mechanisms related to the hyperphosphorylation of Tau protein and the production of beta-amyloid peptide. These are key events leading respectively to the formation of neurofibrillary tangles and senile plaques, which are the neuropathological hallmarks of the disease. Several in vitro and animal studies have shown that the inhibition of GSK3 by lithium and other agents attenuates these pathological processes, reinforcing the notion that GSK3 is a likely target for future disease-modifying therapies for AD. Indeed, a recent study published by our group showed that chronic lithium use is associated with a decrement in the expected prevalence of dementia, in a sample of elderly individuals with bipolar disorder. To investigate this putative neuroprotective effect in a prospective way, the investigators started 24-month randomized, double-blinded controlled trial of lithium for the prevention of dementia in a sample of elderly individuals with amnestic mild cognitive impairment (MCI), a condition associated with increased risk for the development of AD. The clinical and biological outcomes of this trial include the attenuation of cognitive deficits, and the modification of certain biological markers of the disease (as measured in the cerebrospinal fluid, leukocytes and platelets). The objective of the present application is to enable the extension of this ongoing trial to an additional 2-year follow-up. A longer follow-up (48 months) will increase the statistical power to ascertain the primary outcome variables of this study, particularly the con-version from MCI to Alzheimer's disease. This will warrant a more consistent conclusion about the potential of lithium treatment in the prevention of dementia, in addition to a better evaluation of safety and tolerability profiles of the long-term use of lithium in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients with amnestic mild cognitive impairment;
* age: 60 to 80 years-old;

Exclusion Criteria:

* sensory deficiencies that might preclude the administration of cognitive tests;
* active major psychiatry disorder;
* unstable clinical conditions such as cardiac insufficiency, uncontrolled diabetes mellitus, renal failure;
* previous use of lithium salts;
* concurrent participation in other clinical trial or intervention studies;

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
effect of lithium to delay progression of cognitive deficits in patients with amnestic MCI | two year

SECONDARY OUTCOMES:
effect of lithium on CSF levels of Total Tau, Phosphorylated Tau and Amyloid-beta42 | one year
the effect of lithium on the activity of GSK3β in platelets and leukocytes drawn from peripheral blood. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Orestes V Forlenza, Ph.D., Principal Investigator — Department and Institute of Psychiatry, Faculty of Medicine - University of Sao Paulo; Wagner F Gattaz, Ph.D., Study Director — Department and Institute of Psychiatry, Faculty of Medicine - University of Sao Paulo
Locations (1):
- Institute of Psychiatry, Faculty of Medicine - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Forlenza OV, Radanovic M, Talib LL, Gattaz WF. Clinical and biological effects of long-term lithium treatment in older adults with amnestic mild cognitive impairment: randomised clinical trial. Br J Psychiatry. 2019 Nov;215(5):668-674. doi: 10.1192/bjp.2019.76. PMID 30947755
- [Derived] Aprahamian I, Santos FS, dos Santos B, Talib L, Diniz BS, Radanovic M, Gattaz WF, Forlenza OV. Long-term, low-dose lithium treatment does not impair renal function in the elderly: a 2-year randomized, placebo-controlled trial followed by single-blind extension. J Clin Psychiatry. 2014 Jul;75(7):e672-8. doi: 10.4088/JCP.13m08741. PMID 25093483
- [Derived] Forlenza OV, Diniz BS, Radanovic M, Santos FS, Talib LL, Gattaz WF. Disease-modifying properties of long-term lithium treatment for amnestic mild cognitive impairment: randomised controlled trial. Br J Psychiatry. 2011 May;198(5):351-6. doi: 10.1192/bjp.bp.110.080044. PMID 21525519